CLINICAL TRIAL: NCT03743636
Title: Nicotinamide Riboside With and Without Resveratrol to Improve Functioning in Peripheral Artery Disease: The NICE Trial
Brief Title: Nicotinamide Riboside With and Without Resveratrol to Improve Functioning in Peripheral Artery Disease
Acronym: NICE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Mary McDermott, Professor of Medicine at Northwestern University Feinberg School of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU00206660
Record Dates: First submitted 2018-05-20; First posted 2018-11-16 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Peripheral Artery Disease
Keywords: Peripheral Artery Disease; PAD; Resveratrol; Nicotinamide riboside (NR); Six-minute walk; Functional performance
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — nicotinamide-beta-riboside; Resveratrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nicotinamide riboside + resveratrol (Active Comparator): Participants randomized to the NR + resveratrol arm of the study will receive 1,000 mg of NR and 125 mg of resveratrol daily for six months.
  Interventions: Drug: Nicotinamide riboside; Drug: Resveratrol
- Nicotinamide riboside + placebo (Active Comparator): Participants randomized to the NR + placebo arm of the study will receive 1,000 mg of NR and a placebo daily for six months.
  Interventions: Drug: Nicotinamide riboside; Other: Placebo
- Placebo + placebo (Placebo Comparator): Participants randomized to the placebo + placebo arm of study will receive placebo pills.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nicotinamide riboside — Participants randomized to the NR + resveratrol arm or the NR + placebo arm of the study will receive 1,000 mg of NR daily for six months.
  Other Names: NR; Niagen
  Arms: Nicotinamide riboside + placebo; Nicotinamide riboside + resveratrol
Drug: Resveratrol — Participants randomized to the NR + resveratrol arm of the study will receive 125 mg of resveratrol daily for six months.
  Arms: Nicotinamide riboside + resveratrol
Other: Placebo — Participants randomized to the NR + placebo arm of the study will receiving placebo pills that are identical in appearance to resveratrol. Participants randomized to the placebo + placebo arm of the study will receive pills that are identical in appearance to NR and resveratrol. Participants will receive placebo pills daily for six months.
  Arms: Nicotinamide riboside + placebo; Placebo + placebo

SUMMARY:
NICE is a randomized clinical trial that will examine the effects of nicotinamide riboside (NR) both with and without resveratrol to test whether, among people with PAD, NR significantly improves walking performance more than placebo and whether NR combined with resveratrol significantly improves walking performance more than placebo. If findings support the hypotheses, results will be used to design a large, definitive randomized clinical.

The study will randomize 90 participants with PAD to one of the following three groups: NR + resveratrol, NR + placebo, or placebo + placebo.

ELIGIBILITY:
Inclusion Criteria:

All participants will have PAD. PAD will be defined as the following: 1) An ankle-brachial index (ABI) <=0.90 at the baseline study visit or 2) Vascular laboratory evidence or angiographic evidence of PAD. Inclusion based on prior vascular laboratory evidence will be determined by the study principal investigator and includes, for example, a toe brachial index (TBI) < 0.70, Duplex measure showing 70% stenosis or great, a post heel-rise or post-exercise ABI drop of 20% or greater, or ABI values <= 0.90. Angiographic evidence of PAD consists of a stenosis of 70% or greater in a lower extremity artery.

Exclusion Criteria:

1. Above- or below-knee amputation.
2. Critical limb ischemia.
3. Wheelchair-bound or requiring a walker to ambulate.
4. Walking is limited by a symptom other than PAD.
5. Current foot ulcer on bottom of foot.
6. End stage renal disease defined as a GFR less than 20 ml/min/1.73 M2.
7. Significant liver impairment defined as two or more hepatic function enzymes >3.0 times the upper limit of normal. [NOTE: participants who meet this criterion may undergo a re-test of hepatic function tests to determine whether initially elevated hepatic enzymes represented a transient or spurious phenomenon.]
8. Failure to successfully complete the 2-week study run-in.
9. Planned lower extremity revascularization, orthopedic surgery, or other major surgery during the next six months.
10. Lower extremity revascularization, orthopedic surgery, cardiovascular event, coronary revascularization, or other major surgery in the previous three months.
11. Participation in supervised treadmill exercise during the previous three months.
12. Major medical illness including renal disease requiring dialysis, lung disease requiring oxygen, Parkinson's disease, a life-threatening illness with life expectancy less than six months, or cancer requiring treatment in the previous two years. [NOTE: potential participants may still qualify if they have had treatment for an early stage cancer in the past two years and the prognosis is excellent. Participants who only use oxygen at night may still qualify.]
13. Mini-Mental Status Examination (MMSE) score <23 or dementia.
14. Participation in or completion of a clinical trial in the previous three months. [NOTE: after completing a stem cell or gene therapy intervention, participants will become eligible after the final study follow-up visit of the stem cell or gene therapy study so long as at least six months have passed since the final intervention administration. After completing a supplement or drug therapy (other than stem cell or gene therapy), participants will be eligible after the final study follow-up visit as long as at least three months have passed since the final intervention of the trial.]
15. Currently taking a dose of 250 mg or more of nicotinamide riboside, vitamin B3, niacin. Currently taking a slow-release form of niacin. Currently taking resveratrol or has taken any these drug(s) in past six months. Participants taking a multi-vitamin will not be excluded if the dose of vitamin B3 is less than 250 mgs.
16. Increase in angina or angina at rest
17. Non-English speaking.
18. Visual impairment that limits walking ability.
19. Women who are pregnant or who are pre-menopausal will not be eligible.
20. In addition to the above criteria, investigator discretion will be used to determine if the trial is unsafe or not a good fit for the potential participant.

Potentially eligible participants will be advised that Medicare coverage for 12 weeks of supervised treadmill exercise is now available. Potential participants who have not participated in supervised treadmill exercise covered by Medicare and who desire to participate will be referred back to their physician for follow-up. These individuals may become eligible six months after they complete supervised treadmill exercise.

Vulnerable populations (fetuses, pregnant women, children, prisoners, and institutionalized persons) and adults unable to consent will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary M McDermott, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nayak P, Polonsky T, Tian L, Greenland P, Xu S, Zhang D, Zhao L, Criqui MH, Kibbe MR, Gladders B, Goodney P, Ho K, Guralnik JM, McDermott MM. Medical therapies, comorbid conditions, and functional performance in people with peripheral artery disease enrolled in clinical trials between 2004 and 2021. Vasc Med. 2023 Apr;28(2):144-146. doi: 10.1177/1358863X221145533. Epub 2023 Jan 1. PMID 36588397

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Started | 33 | 28 | 29
3-month Follow-up | 30 | 26 | 27
Completed | 33 | 28 | 29
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo | Total
Number analyzed (Participants) | 33 | 28 | 29 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.73 (8.97) | 73.21 (9.97) | 69.72 (8.29) | 71.18 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 16 | 42
  Male | 19 | 16 | 13 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 31 | 25 | 27 | 83
  Unknown or Not Reported | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 19 | 8 | 16 | 43
  White | 13 | 19 | 12 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Ankle brachial index [Mean (Standard Deviation); unit: ratio] — The ABI test compares the blood pressures in the arms and legs to measure the blood flow to the legs. A lower ABI would indicate the narrowing or blockage of leg arteries.
  The Ankle Brachial Index is a ratio of Doppler recorded pressures in the lower and upper extremities. The normal range for ABI is 1.10-1.40. Peripheral artery disease is defined as an ABI < 0.90.
  ABI is calculated by dividing the average of the lower extremity arterial pressures (dorsalis pedis and posterior tibial pressures) by the average of the systolic brachial pressures.
  ratio | 0.67 (0.20) | 0.72 (0.18) | 0.64 (0.18) | 0.68 (0.19)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29.30 (6.66) | 28.65 (3.61) | 30.37 (6.39) | 29.44 (5.76)
6-min walk distance [Mean (Standard Deviation); unit: meters] | 336.61 (80.75) | 339.18 (103.07) | 325.60 (112.51) | 333.86 (97.90)

OUTCOME MEASURES:

1. Primary Outcome: Six-minute Walk Distance (NR Alone vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR alone improves six-minute walk distance at 6-month follow-up, compared to placebo.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 29
meters | -6.93 (7.84) | 7.00 (8.69) | -10.58 (8.45)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Placebo vs Placebo + Placebo; Test type: Superiority; p = 0.0775, Mixed Models Analysis; Mean Difference (Final Values) = 17.57, 90% CI 1-sided [lower limit 1.77]

2. Primary Outcome: Six-minute Walk Distance (NR/Resveratrol vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves six-minute walk performance at 6-month follow-up, compared to placebo.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 29
meters | -6.93 (7.84) | 7.00 (8.69) | -10.58 (8.45)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Placebo + Placebo; Test type: Superiority; p = 0.3762, Mixed Models Analysis; Mean Difference (Final Values) = 3.65, 90% CI 1-sided [lower limit -11.24]

3. Secondary Outcome: Six-minute Walk Distance (NR Alone vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR alone improves six-minute walk performance at 3-month follow-up, compared to placebo.
Time Frame: Baseline to 3-month follow-up
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 29
meters | 2.99 (7.67) | 4.78 (8.28) | -17.64 (8.03)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Placebo vs Placebo + Placebo; Test type: Superiority; p = 0.0294, Mixed Models Analysis; Mean Difference (Final Values) = 22.42, 90% CI 1-sided [lower limit 7.31]

4. Secondary Outcome: Six-minute Walk Distance (NR/Resveratrol vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves six-minute walk performance at 3-month follow-up, compared to placebo.
Time Frame: Baseline to 3-month follow-up
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 29
meters | 2.99 (7.67) | 4.78 (8.28) | -17.64 (8.03)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Placebo + Placebo; Test type: Superiority; p = 0.0336, Mixed Models Analysis; Mean Difference (Final Values) = 20.63, 90% CI 1-sided [lower limit 6.26]

5. Secondary Outcome: Six-minute Walk Distance (NR/Resveratrol vs. NR Alone)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves six-minute walk performance at 3-month follow-up, compared to NR alone.
Time Frame: Baseline to 3-month follow-up
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 29
meters | 2.99 (7.67) | 4.78 (8.28) | -17.64 (8.03)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Nicotinamide Riboside + Placebo; Test type: Superiority; p = 0.5620, Mixed Models Analysis; Mean Difference (Final Values) = -1.78, 90% CI 1-sided [lower limit -16.51]

6. Secondary Outcome: Six-minute Walk Distance (NR/Resveratrol vs. NR Alone)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves six-minute walk performance at 6-month follow-up, compared to NR alone.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 29
meters | -6.93 (7.84) | 7.00 (8.69) | -10.58 (8.45)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Nicotinamide Riboside + Placebo; Test type: Superiority; p = 0.8797, Mixed Models Analysis; Mean Difference (Final Values) = -13.93, 90% CI 1-sided [lower limit -29.15]

7. Secondary Outcome: Maximal Treadmill Walking Time (NR Alone vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR alone improves maximal treadmill walking time at 6-month follow-up, compared to placebo.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 8 | 10 | 8
minutes | 0.57 (1.11) | 0.89 (0.94) | -1.17 (0.97)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Placebo vs Placebo + Placebo; Test type: Superiority; p = 0.0752, ANCOVA; Mean Difference (Final Values) = 2.06, 90% CI 1-sided [lower limit 0.24]

8. Secondary Outcome: Walking Impairment Questionnaire (WIQ) Distance Score (NR Alone vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR alone improves the Walking Impairment Questionnaire (WIQ) distance score at 6-month follow-up, compared to placebo.
  The WIQ is a well validated questionnaire that measures patient-reported walking limitations in distance and speed and stair-climbing. They are scored on a 0-100 scale and that 100 indicates the best possible score.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 28
score on a scale | 0.82 (3.96) | -1.24 (4.42) | 5.86 (4.31)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Placebo vs Placebo + Placebo; Test type: Superiority; p = 0.8703, ANCOVA; Mean Difference (Final Values) = -7.10, 90% CI 1-sided [lower limit -15.19]

9. Secondary Outcome: Physical Activity (NR Alone vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR alone improves physical activity at 6-month follow-up, compared to placebo.
  The physical activity outcome was measured with the ActiGraph, in Activity Units. Higher scores indicate greater activity. The lowest possible score is zero, indicating sedentary time.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Activity count per day
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 28 | 25 | 25
Activity count per day | -7743 (6478) | 4094 (7109) | -6901 (6889)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Placebo vs Placebo + Placebo; Test type: Superiority; p = 0.1402, ANCOVA; Mean Difference (Final Values) = 10995, 90% CI 1-sided [lower limit -2078]

10. Secondary Outcome: Maximal Treadmill Walking Time (NR/Resveratrol vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves maximal treadmill walking time at 6-month follow-up, compared to placebo.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 8 | 10 | 8
minutes | 0.57 (1.11) | 0.89 (0.94) | -1.17 (0.97)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Placebo + Placebo; Test type: Superiority; p = 0.1249, ANCOVA; Mean Difference (Final Values) = 1.74, 90% CI 1-sided [lower limit -0.21]

11. Secondary Outcome: Walking Impairment Questionnaire (WIQ) Distance Score (NR/Resveratrol vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves the Walking Impairment Questionnaire distance score at 6-month follow-up, compared to placebo.
  The WIQ is a well validated questionnaire that measures patient-reported walking limitations in distance and speed and stair-climbing. They are scored on a 0-100 scale and that 100 indicates the best possible score.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 28
score on a scale | 0.82 (3.96) | -1.24 (4.42) | 5.86 (4.31)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Placebo + Placebo; Test type: Superiority; p = 0.8039, ANCOVA; Mean Difference (Final Values) = -5.05, 90% CI 1-sided [lower limit -12.62]

12. Secondary Outcome: Physical Activity (NR/Resveratrol vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves physical activity at 6-month follow-up, compared to placebo.
  The physical activity outcome was measured with the ActiGraph, in Activity Units. Higher scores indicate greater activity. The lowest possible score is zero, indicating sedentary time.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Activity count per day
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 28 | 25 | 25
Activity count per day | -7743 (6478) | 4094 (7109) | -6901 (6889)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Placebo + Placebo; Test type: Superiority; p = 0.5352, ANCOVA; Mean Difference (Final Values) = -842, 90% CI 1-sided [lower limit -13125]

13. Secondary Outcome: Maximal Treadmill Walking Time (NR/Resveratrol vs. NR Alone)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves maximal treadmill walking time at 6-month follow-up, compared to NR alone.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 8 | 10 | 8
minutes | 0.57 (1.11) | 0.89 (0.94) | -1.17 (0.97)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Nicotinamide Riboside + Placebo; Test type: Superiority; p = 0.5777, ANCOVA; Mean Difference (Final Values) = -0.32, 90% CI 1-sided [lower limit -2.46]

14. Secondary Outcome: Walking Impairment Questionnaire (WIQ) Distance Score (NR/Resveratrol vs. NR Alone)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves the Walking Impairment Questionnaire (WIQ) distance score at 6-month follow-up, compared to NR alone.
  The WIQ is a well validated questionnaire that measures patient-reported walking limitations in distance and speed and stair-climbing. They are scored on a 0-100 scale and that 100 indicates the best possible score.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 28
score on a scale | 0.82 (3.96) | -1.24 (4.42) | 5.86 (4.31)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Nicotinamide Riboside + Placebo; Test type: Superiority; p = 0.3662, ANCOVA; Mean Difference (Final Values) = 2.06, 90% CI 1-sided [lower limit -5.69]

15. Secondary Outcome: Physical Activity (NR/Resveratrol vs. NR Alone)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves physical activity at 6-month follow-up, compared to NR alone..
  The physical activity outcome was measured with the ActiGraph, in Activity Units. Higher scores indicate greater activity. The lowest possible score is zero, indicating sedentary time.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Activity count per day
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 28 | 25 | 25
Activity count per day | -7743 (6478) | 4094 (7109) | -6901 (6889)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Nicotinamide Riboside + Placebo; Test type: Superiority; p = 0.8866, ANCOVA; Mean Difference (Final Values) = -11837, 90% CI 1-sided [lower limit -24396]

16. Secondary Outcome: Six-minute Walk Distance (NR/Resveratrol or NR Alone vs. Placebo)
Description: Participants with PAD who received NR alone and those who received NR + resveratrol will be combined into one group and compared to the group receiving placebo, to determine whether NR alone or NR+ resveratrol (combined group)have greater improvement in six-minute walk distance, compared to those randomized to placebo.
  Mixed model for repeated measures is applied to Placebo vs. 2 NR groups combined. The reported results of within group change and between group difference are Least Squares Mean (Standard Error) from the model adjusted for baseline six-minute walk + age + sex + race + resveratrol usage.
Time Frame: Baseline to 3-month follow-up
Measure: Least Squares Mean (Standard Error); unit: meters
Groups:
- Two NR Groups Combined: NR+Resveratrol and NR alone groups combined
Arm/Group | Placebo + Placebo | Two NR Groups Combined
Number analyzed (Participants) | 29 | 61
meters | -21.34 (9.66) | 3.92 (5.61)
Statistical Analysis 1: Comparison: Placebo + Placebo vs Two NR Groups Combined; Mixed models for repeated measures were used to compare 3-month change in 6MW distance between the NR/resveratrol vs placebo groups and between the NR alone vs placebo groups using baseline, 3-month, and 6-month values, adjusted for age, sex, race, and baseline 6MW; Test type: Superiority — Mixed model for repeated measures is applied to Placebo vs. 2 NR groups combined. The reported results of within group change and between group difference are Least Squares Mean (Standard Error) from the model adjusted for baseline six-minute walk + age + sex + race + resveratrol usage; p = 0.0153, Mixed Models Analysis — The a priori statistical analysis plan defined a one-sided P value of < 0.10 to define statistical significance; Mean Difference (Final Values) = 25.25, 90% CI 1-sided [lower limit 10.43]

17. Secondary Outcome: Six-minute Walk Distance (NR/Resveratrol or NR Alone vs. Placebo)
Description: as for outcome 16
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: meters
Arm/Group | Placebo + Placebo | Two NR Groups Combined
Number analyzed (Participants) | 29 | 61
meters | -14.29 (9.97) | -0.24 (5.81)
Statistical Analysis 1: Comparison: Placebo + Placebo vs Two NR Groups Combined; Mixed models for repeated measures were used to compare 6-month change in 6MW distance between the NR/resveratrol vs placebo groups and between the NR alone vs placebo groups using baseline, 3-month, and 6-month values, adjusted for age, sex, race, and baseline 6MW; Test type: Superiority — [test comment as in outcome 16, analysis 1]; p = 0.1195, Mixed Models Analysis; Mean Difference (Final Values) = 14.05, 90% CI 1-sided [lower limit -1.25]

18. Secondary Outcome: Maximal Treadmill Walking Time (NR/Resveratrol or NR Alone vs. Placebo)
Description: Participants with PAD who received NR alone and those who received NR + resveratrol will be combined into one group and compared to the group receiving placebo, to determine whether NR alone or NR+ resveratrol (combined group)have greater improvement in maximal treadmill walking time, compared to those randomized to placebo.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo + Placebo | Two NR Groups Combined
Number analyzed (Participants) | 8 | 18
minutes | -1.33 (1.28) | 0.73 (0.64)
Statistical Analysis 1: Comparison: Placebo + Placebo vs Two NR Groups Combined; Mixed model for repeated measures is applied to Placebo vs. 2 NR groups combined. The reported results of within group change and between group difference are Least Squares Mean (Standard Error) from the model adjusted for baseline six-minute walk + age + sex + race + resveratrol usage; Test type: Superiority; p = 0.0752, ANCOVA — The a priori statistical analysis plan defined a one-sided P value of < 0.10 to define statistical significance; Mean Difference (Final Values) = 2.06, 90% CI 1-sided [lower limit 0.24]

19. Secondary Outcome: Walking Impairment Questionnaire (WIQ) Distance Score (NR/Resveratrol or NR Alone vs. Placebo)
Description: Participants with PAD who received NR alone and those who received NR + resveratrol will be combined into one group and compared to the group receiving placebo, to determine whether NR alone or NR+ resveratrol (combined group)have greater improvement in Walking Impairment Questionnaire distance score, compared to those randomized to placebo.
  The WIQ is a well validated questionnaire that measures patient-reported walking limitations in distance and speed and stair-climbing. They are scored on a 0-100 scale and that 100 indicates the best possible score.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Placebo | Two NR Groups Combined
Number analyzed (Participants) | 28 | 61
score on a scale | 6.89 (5.29) | -0.21 (2.94)
Statistical Analysis 1: Comparison: Placebo + Placebo vs Two NR Groups Combined; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.8703, ANCOVA; Mean Difference (Final Values) = -7.10, 90% CI 1-sided [lower limit -15.19]

20. Secondary Outcome: Physical Activity (NR/Resveratrol or NR Alone vs. Placebo)
Description: Participants with PAD who received NR alone and those who received NR + resveratrol will be combined into one group and compared to the group receiving placebo, to determine whether NR alone or NR+ resveratrol (combined group)have greater improvement in physical activity, compared to those randomized to placebo.
  The physical activity outcome was measured with the ActiGraph, in Activity Units. Higher scores indicate greater activity. The lowest possible score is zero, indicating sedentary time.
  Mixed model for repeated measures is applied to Placebo vs. 2 NR groups combined. The reported results of within group change and between group difference are Least Squares Mean (Standard Error) from the model adjusted for baseline six-minute walk + age + sex + race + resveratrol usage.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Activity count per day
Arm/Group | Placebo + Placebo | Two NR Groups Combined
Number analyzed (Participants) | 25 | 53
Activity count per day | -12819 (8528) | -1824 (4763)
Statistical Analysis 1: Comparison: Placebo + Placebo vs Two NR Groups Combined; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.1402, ANCOVA; Mean Difference (Final Values) = 10995, 90% CI 1-sided [lower limit -2078]

21. Secondary Outcome: NAD+ Abundance in Gastrocnemius Muscle (NR/Resveratrol or NR Alone vs. Placebo)
Description: The outcome measure is the comparison of 6-month change in gastrocnemius muscle biopsy measures of NAD+ abundance between NR and placebo and between NR + resveratrol and placebo. Participants with PAD who received NR alone and those who received NR + resveratrol will be combined into one group and compared to the group receiving placebo, to determine whether NR alone or NR+ resveratrol (combined group) have greater improvement in NAD+ abundance, compared to those randomized to placebo. Measurements of NAD+ abundance were completed using High Performance Liquid Chromatography (HPLC) with a Shimadzu LC-20A pump and UV-VIS detector using a Supelco LC-18-Tcolumn, normalized to muscle weight.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: pmol/mg
Arm/Group | Placebo + Placebo | Two NR Groups Combined
Number analyzed (Participants) | 5 | 12
pmol/mg | 43.83 (26.15) | 8.70 (17.92)
Statistical Analysis 1: Comparison: Placebo + Placebo vs Two NR Groups Combined; Test type: Superiority; p = 0.8401, ANCOVA; Mean Difference (Final Values) = -35.13, 90% CI 1-sided [lower limit -81.20]

22. Secondary Outcome: Satellite Cell Abundance in Gastrocnemius Muscle (NR/Resveratrol or NR Alone vs. Placebo)
Description: The outcome measure is the comparison of 6-month changes in gastrocnemius muscle biopsy measures of satellite cell abundance between NR and placebo and between NR + resveratrol and placebo. Participants with PAD who received NR alone and those who received NR + resveratrol will be combined into one group and compared to the group receiving placebo, to determine whether NR alone or NR+ resveratrol (combined group) have greater improvement in satellite cell abundance, compared to those randomized to placebo. Satellite cell abundance was measured via density (satellite cells/100 fibers) using antibodies against: Pax7, type 1 myosin, and laminin.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: satellite cells/100 fibers
Arm/Group | Placebo + Placebo | Two NR Groups Combined
Number analyzed (Participants) | 5 | 11
satellite cells/100 fibers | -11.95 (5.18) | -0.81 (3.32)
Statistical Analysis 1: Comparison: Placebo + Placebo vs Two NR Groups Combined; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.0602, ANCOVA; Mean Difference (Final Values) = 11.14, 90% CI 1-sided [lower limit 2.16]

23. Secondary Outcome: Gastrocnemius Muscle Fiber Phenotype(NR/Resveratrol or NR Alone vs. Placebo)
Description: The outcome measure is the comparison of 6-month changes in gastrocnemius muscle biopsy measures of Percent Type 1 myofibers (%) between NR and placebo and between NR + resveratrol and placebo. Participants with PAD who received NR alone and those who received NR + resveratrol will be combined into one group and compared to the group receiving placebo, to determine whether NR alone or NR+ resveratrol (combined group) have greater improvement in muscle fiber phenotype, compared to those randomized to placebo. Measurements of fiber type % were determined on frozen muscle sections using antibodies against: Pax7, type 1 myosin, and laminin.
  Mixed model for repeated measures is applied to Placebo vs. 2 NR groups combined. The reported results of within group change and between group difference are Least Squares Mean (Standard Error) from the model adjusted for baseline six-minute walk + age + sex + race + resveratrol usage.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Placebo + Placebo | Two NR Groups Combined
Number analyzed (Participants) | 5 | 11
percentage | -2.88 (3.58) | -8.09 (5.75)
Statistical Analysis 1: Comparison: Placebo + Placebo vs Two NR Groups Combined; Test type: Superiority; p = 0.2378, ANCOVA; Mean Difference (Final Values) = 5.21, 90% CI 1-sided [lower limit -4.47]

24. Other Pre Specified Outcome: Gastrocnemius Muscle Satellite Cell Abundance (NR/Resveratrol vs. Placebo and NR vs. Placebo)
Description: Investigators will perform calf muscle biopsies to determine whether among participants with PAD, those randomized to NR + resveratrol and NR alone have increased satellite cell abundance compared to the placebo group. Satellite cell abundance was measured via density (satellite cells/100 fibers) using antibodies against: Pax7, type 1 myosin, and laminin.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: satellite cells/100 fibers
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 4 | 7 | 5
satellite cells/100 fibers | -3.36 (4.33) | 1.73 (4.52) | -9.41 (3.80)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Placebo + Placebo; Mixed model for repeated measures is applied to 3 groups comparisons. The reported results of within group change and between group difference are Least Squares Mean (Standard Error) from the model adjusted for baseline six-minute walk + age + sex + race + resveratrol usage; Test type: Superiority; p = 0.1589, ANCOVA; Mean Difference (Final Values) = 6.05, 90% CI 1-sided [lower limit -1.86]
Statistical Analysis 2: Comparison: Nicotinamide Riboside + Placebo vs Placebo + Placebo; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.0602, ANCOVA; Mean Difference (Final Values) = 11.14, 90% CI 1-sided [lower limit 2.16]

25. Other Pre Specified Outcome: NAD+ Abundance in Gastrocnemius Muscle (NR/Resveratrol vs. Placebo and NR vs. Placebo)
Description: Investigators will perform calf muscle biopsies to determine whether among participants with PAD, those randomized to NR + resveratrol and NR alone have increased calf muscle NAD+ abundance, compared to the placebo group. Measurements of NAD+ abundance were completed using High Performance Liquid Chromatography (HPLC) with a Shimadzu LC-20A pump and UV-VIS detector using a Supelco LC-18-Tcolumn, normalized to muscle weight.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: pmol/mg
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 5 | 7 | 5
pmol/mg | 31.39 (22.57) | -13.99 (23.44) | 21.14 (20.03)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Placebo + Placebo; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.3724, ANCOVA; Mean Difference (Final Values) = 10.25, 90% CI 1-sided [lower limit -31.79]
Statistical Analysis 2: Comparison: Nicotinamide Riboside + Placebo vs Placebo + Placebo; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.8401, ANCOVA; Mean Difference (Final Values) = -35.13, 90% CI 1-sided [lower limit -81.20]

26. Other Pre Specified Outcome: Muscle Fiber Phenotype in Gastrocnemius Muscle (NR/Resveratrol vs. Placebo and NR vs. Placebo)
Description: Investigators will perform calf muscle biopsies to determine whether among participants with PAD, those randomized to NR + resveratrol and NR alone have improved muscle fiber phenotype (Percent Type 1 myofibers (%)), compared to the placebo group. Measurements of fiber type % were determined on frozen muscle sections using antibodies against: Pax7, type 1 myosin, and laminin.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 4 | 7 | 5
percentage | -5.94 (4.88) | 0.17 (4.86) | -5.04 (4.12)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Placebo + Placebo; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.5558, ANCOVA; Mean Difference (Final Values) = -0.90, 90% CI 1-sided [lower limit -9.52]
Statistical Analysis 2: Comparison: Nicotinamide Riboside + Placebo vs Placebo + Placebo; [analysis description as in outcome 24, analysis 1]; Test type: Superiority; p = 0.2378, ANCOVA; Mean Difference (Final Values) = 5.21, 90% CI 1-sided [lower limit -4.47]

27. Other Pre Specified Outcome: Walking Impairment Questionnaire (WIQ) Speed Score (NR Alone vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR alone improves the Walking Impairment Questionnaire speed and stair climbing score at 6-month follow-up, compared to placebo.
  The WIQ is a well validated questionnaire that measures patient-reported walking limitations in distance and speed and stair-climbing. They are scored on a 0-100 scale and that 100 indicates the best possible score.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 28
score on a scale | -0.82 (3.08) | 0.22 (3.43) | 2.93 (3.34)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Placebo vs Placebo + Placebo; Test type: Superiority; p = 0.7112, ANCOVA; Mean Difference (Final Values) = -2.71, 90% CI 1-sided [lower limit -8.97]

28. Other Pre Specified Outcome: Short-Form Physical Functioning (SF-36) Score (NR Alone vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR alone improves the Walking Impairment Questionnaire speed and stair climbing scores and the Short-Form Physical Functioning score at 6-month follow-up, compared to placebo.
  The SF-36 measures health status. The score range is 0-100, where 100 is best.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 28
score on a scale | 0.65 (2.89) | -3.40 (3.23) | 4.00 (3.15)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Placebo vs Placebo + Placebo; Test type: Superiority; p = 0.9449, ANCOVA; Mean Difference (Final Values) = -7.40, 90% CI 1-sided [lower limit -13.31]

29. Other Pre Specified Outcome: Walking Impairment Questionnaire (WIQ) Stair Climbing Score (NR/Resveratrol vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves the Walking Impairment Questionnaire speed and stair climbing scores at 6-month follow-up, compared to placebo.
  The WIQ is a well validated questionnaire that measures patient-reported walking limitations in distance and speed and stair-climbing. They are scored on a 0-100 scale and that 100 indicates the best possible score.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 28
score on a scale | -2.64 (3.18) | 2.09 (3.55) | -2.15 (3.46)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Placebo + Placebo; Test type: Superiority; p = 0.5409, ANCOVA; Mean Difference (Final Values) = -0.48, 90% CI 1-sided [lower limit -6.57]

30. Other Pre Specified Outcome: Short-Form Physical Functioning (SF-36) Score (NR/Resveratrol vs. Placebo)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves the Short-Form Physical Functioning score at 6-month follow-up, compared to placebo.
  The SF-36 measures health status. The score range is 0-100, where 100 is best.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 28
score on a scale | 0.65 (2.89) | -3.40 (3.23) | 4.00 (3.15)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Placebo + Placebo; Test type: Superiority; p = 0.7814, ANCOVA; Mean Difference (Final Values) = -3.35, 90% CI 1-sided [lower limit -8.89]

31. Other Pre Specified Outcome: Walking Impairment Questionnaire (WIQ) Speed Score (NR/Resveratrol vs. NR Alone)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves the Walking Impairment Questionnaire speed and stair climbing score at 6-month follow-up, compared to NR alone.
  The WIQ is a well validated questionnaire that measures patient-reported walking limitations in distance and speed and stair-climbing. They are scored on a 0-100 scale and that 100 indicates the best possible score.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 28
score on a scale | -0.82 (3.08) | 0.22 (3.43) | 2.93 (3.34)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Nicotinamide Riboside + Placebo; Test type: Superiority; p = 0.5884, ANCOVA; Mean Difference (Final Values) = -1.04, 90% CI 1-sided [lower limit -7.07]

32. Other Pre Specified Outcome: Short-Form Physical Functioning (SF-36) Score (NR/Resveratrol vs. NR Alone)
Description: Among participants with PAD, investigators will determine whether NR combined with resveratrol improves the Walking Impairment Questionnaire speed and stair climbing scores and the Short-Form Physical Functioning score at 6-month follow-up, compared to NR alone.
  The SF-36 measures health status. The score range is 0-100, where 100 is best.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
Number analyzed (Participants) | 33 | 28 | 28
score on a scale | 0.65 (2.89) | -3.40 (3.23) | 4.00 (3.15)
Statistical Analysis 1: Comparison: Nicotinamide Riboside + Resveratrol vs Nicotinamide Riboside + Placebo; Test type: Superiority; p = 0.1787, ANCOVA; Mean Difference (Final Values) = 4.05, 90% CI 1-sided [lower limit -1.60]

33. Other Pre Specified Outcome: Walking Impairment Questionnaire (WIQ) Speed Score (NR/Resveratrol or NR Alone vs. Placebo)
Description: Participants with PAD who received NR alone and those who received NR + resveratrol will be combined into one group and compared to the group receiving placebo, to determine whether NR alone or NR+ resveratrol (combined group) have greater improvement in the Walking Impairment Questionnaire (WIQ) speed and stair climbing score at 6-month follow-up, compared to placebo.
  The WIQ is a well validated questionnaire that measures patient-reported walking limitations in distance and speed and stair-climbing. They are scored on a 0-100 scale and that 100 indicates the best possible score.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Placebo | Two NR Groups Combined
Number analyzed (Participants) | 28 | 61
score on a scale | 2.41 (4.10) | -0.30 (2.28)
Statistical Analysis 1: Comparison: Placebo + Placebo vs Two NR Groups Combined; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.7112, ANCOVA; Mean Difference (Final Values) = -2.71, 90% CI 1-sided [lower limit -8.97]

34. Other Pre Specified Outcome: Short-Form Physical Functioning (SF-36) Score (NR/Resveratrol or NR Alone vs. Placebo)
Description: Participants with PAD who received NR alone and those who received NR + resveratrol will be combined into one group and compared to the group receiving placebo, to determine whether NR alone or NR+ resveratrol (combined group) have greater improvement in the Short-Form Physical Functioning score at 6-month follow-up, compared to placebo.
  The SF-36 measures health status. The score range is 0-100, where 100 is best.
Time Frame: Baseline to 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo + Placebo | Two NR Groups Combined
Number analyzed (Participants) | 28 | 61
score on a scale | 6.02 (3.87) | -1.37 (2.15)
Statistical Analysis 1: Comparison: Placebo + Placebo vs Two NR Groups Combined; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.9449, ANCOVA; Mean Difference (Final Values) = -7.40, 90% CI 1-sided [lower limit -13.31]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected monthly from baseline to 6-month follow-up.
Arm/Group | Nicotinamide Riboside + Resveratrol | Nicotinamide Riboside + Placebo | Placebo + Placebo
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/28 | 0/29
Serious Adverse Events (participants affected / at risk) | 9/33 | 6/28 | 6/29
Other Adverse Events (participants affected / at risk) | 24/33 | 18/28 | 21/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotinamide Riboside + Resveratrol (N=33) | Nicotinamide Riboside + Placebo (N=28) | Placebo + Placebo (N=29)
Lower extremity revascularization (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (General disorders) | 1 (1) | 1 (1) | 1 (2)
Hypertension (General disorders) | 1 (1) | 0 (0) | 1 (1)
Coronary revascularization (General disorders) | 0 (0) | 0 (0) | 1 (1)
Carotid endarterectomy (General disorders) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (General disorders) | 0 (0) | 1 (1) | 0 (0)
Stroke (General disorders) | 2 (2) | 0 (0) | 0 (0)
Coronary ischemia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (General disorders) | 1 (1) | 1 (1) | 0 (0)
Lightheadedness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (General disorders) | 0 (0) | 0 (0) | 1 (1)
Mass in groin region (General disorders) | 0 (0) | 1 (1) | 0 (0)
Opioid withdrawal (General disorders) | 1 (1) | 0 (0) | 0 (0)
COPD (General disorders) | 0 (0) | 1 (1) | 0 (0)
Jaw pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Angina (General disorders) | 0 (0) | 0 (0) | 1 (1)
TIA (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Lung biopsy (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotinamide Riboside + Resveratrol (N=33) | Nicotinamide Riboside + Placebo (N=28) | Placebo + Placebo (N=29)
Nausea or vomiting (General disorders) | 12 (18) | 4 (9) | 7 (8)
Diarrhea (General disorders) | 18 (33) | 11 (20) | 8 (19)
Abdominal discomfort (General disorders) | 13 (21) | 11 (22) | 13 (26)
Flushing (General disorders) | 9 (26) | 9 (16) | 10 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/36/NCT03743636/Prot_SAP_000.pdf